CLINICAL TRIAL: NCT00003735
Title: A Phase II Study of Oral Topotecan in Children With Relapsed Acute Leukemia
Brief Title: Chemotherapy in Treating Children With Relapsed Acute Leukemia, Acute Myeloid Leukemia, or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09714; CCG-09714; CDR0000066850; COG-09714 (Other: Children's Oncology Group)
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; blastic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Topotecan

ARMS (2):
- Stratum 1 - Stage 1 (Experimental): Topotecan hydrochloride (0.8 mg/m²/day) by mouth for 21 days. Bone marrow will be obtained on approximately Day 28 of Course 1 and 2 and in any course where the CBC suggests that a relapse has occurred. One additional course may be given if the blood is cleared of blasts and the bone marrow is M1, M2 or M3. The patient is off protocol therapy if blasts are still present in the blood and the marrow is M3. Subsequent courses of topotecan may be given only if the bone marrow after Course 2 is M1 or M2. If the bone marrow is M2 on Day 28 of any course, another bone marrow aspirate will be done at the end of the next course. If the patient is in CR, a bone marrow aspirate will be required only every other course unless the peripheral blood suggests that a relapse has occurred. Each subsequent course should begin within six weeks of the start of the previous course.
  Interventions: Drug: topotecan hydrochloride
- Stratum 2 - Stage 2 (Experimental): Topotecan hydrochloride (0.8 mg/m²/day) by mouth for 21 days. Bone marrow will be obtained on approximately Day 28 of Course 1 and 2 and in any course where the CBC suggests that a relapse has occurred. One additional course may be given if the blood is cleared of blasts and the bone marrow is M1, M2 or M3. The patient is off protocol therapy if blasts are still present in the blood and the marrow is M3. Subsequent courses of topotecan may be given only if the bone marrow after Course 2 is M1 or M2. If the bone marrow is M2 on Day 28 of any course, another bone marrow aspirate will be done at the end of the next course. If the patient is in CR, a bone marrow aspirate will be required only every other course unless the peripheral blood suggests that a relapse has occurred. Each subsequent course should begin within six weeks of the start of the previous course.
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride — given by mouth
  Other Names: Hycamptamine; SK&B 104864-A; 9-dimethylaminomethyl-10-hydroxycamptothecin hydrochloride; IND #56, 270.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of topotecan in treating children who have relapsed acute leukemia, acute myeloid leukemia, or blast phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with relapsed acute lymphocytic leukemia, acute myeloid leukemia, or blastic phase chronic myelogenous leukemia treated with oral topotecan. II. Determine the toxic effects and pharmacokinetics of this regimen in these patients.

OUTLINE: Patients are stratified by disease type (acute lymphocytic leukemia vs acute myeloid leukemia). Patients receive oral topotecan once daily on days 1-21. Courses repeat every 28 days in the absence of blasts in the blood, M3 bone marrow, or unacceptable toxicity. Patients are followed every 6 months until death.

PROJECTED ACCRUAL: A total of 50 patients (25 per stratum) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven relapsed acute lymphocytic leukemia, acute myeloid leukemia, or blastic phase chronic myelogenous leukemia Refractory to conventional therapy and other therapies of higher priority May have concurrent extramedullary relapse except for testicular relapse or other extramedullary sites that may require concurrent radiotherapy

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 times normal SGOT or SGPT less than 5 times normal Renal: Creatinine no greater than 1.5 times normal Other: Able to take oral liquid medication No GI neuropathy No other condition that may affect absorption of drug No diabetes mellitus Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior bone marrow transplantation (BMT) or peripheral blood stem cell transplantation (PBSCT) allowed and recovered At least 2 weeks since prior cytokine therapy and recovered No concurrent immune modulator therapy No concurrent cytokines including interleukin-11, interleukin-2, and epoetin alfa Chemotherapy: At least 2 weeks since prior chemotherapy (4 weeks for nitrosoureas) and recovered No more than 3 prior chemotherapy regimens No other concurrent chemotherapy Endocrine therapy: No concurrent steroids Radiotherapy: No prior craniospinal radiotherapy Prior total body irradiation allowed as part of BMT or PBSCT and recovered Concurrent radiotherapy for localized painful lesions allowed Surgery: Not specified Other: No concurrent metoclopramide or cisapride to maintain motility or gastric emptying No concurrent H2 antagonists No concurrent proton pump inhibitors No concurrent antacids for gastritis, gastroesophageal reflux, or ulcers (gastric or duodenal) No antacid therapy for 6 hours before and for 90 minutes after topotecan administration

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 1998-12; Primary Completion 2002-11 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 21 days
  For each stratum, this trial will determine topotecan to have insufficient activity for further investigation with probability 0.10 if the true response rate is 20%. For each stratum, this trial will determine topotecan to be of sufficient activity to warrant further investigation with probability 0.12 if the true response rate is 5%. Any patient who receives at least 21 days of therapy will be considered evaluable for response.

CONTACTS AND LOCATIONS:
Overall Officials: John S. Holcenberg, MD, Study Chair — Seattle Children's Hospital
Locations (38):
- United States (35):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia